CLINICAL TRIAL: NCT01245777
Title: Exploratory Study of the Efficacy, Practicability and Safety of Intravenous Iron Supplementation Therapy in Moderate to Severe Restless Legs Syndrome With Iron Deficiency or Anaemia in the 3rd Trimester of Pregnancy
Brief Title: Restless Legs Syndrome With Iron Deficiency or Anaemia in the 3rd Trimester of Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITiRiP-1
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Restless Leg Syndrome; Iron Deficiency Anemia
Keywords: RLS; Pregnancy; Iron Deficiency; Anaemia
MeSH Terms: conditions — Restless Legs Syndrome; Anemia, Iron-Deficiency; Iron Deficiencies; Anemia | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ferric carboxymaltose (Experimental): Hb> 11 g/dl and Ferritin < 35 (controlled by CRP): 500mg to correct iron deficiency Hb ≥ 10 and < 11g/dl; Ferritin < 35 (controlled by CRP): 700 mg Hb ≥9 and < 10 g/dl; Ferritin < 35 (controlled by CRP): 800 mg Hb < 9g/dl; Ferritin < 35 (controlled by CRP): 900 mg
  Interventions: Drug: ferric carboxymaltose

INTERVENTIONS:
Drug: ferric carboxymaltose — 20 women with Restless Legs Syndrome (RLS) and iron deficiency and/ or anaemia in the third trimester of pregnancy will receive intravenous Ferric carboxymaltose in one or two single doses.
  Other Names: Ferinject

SUMMARY:
In pregnancy Restless Legs Syndrome(RLS) is more common than in the general population. During pregnancy iron tablets are the only available safe medication but their efficacy is rather poor. It is the aim of this study to examine the efficacy, practicability and safety of the drug Ferinject® containing the active agent Ferric carboxymaltose for the therapy of Restless Legs Syndrome(RLS) during pregnancy in the case of iron deficiency or anaemia.

20 women with RLS and iron deficiency and/ or anaemia in the third trimester of pregnancy will receive intravenous Ferric carboxymaltose in one or two single doses. Repeated blood tests, pre-and post-therapy actigraphy as well as repeated answering of questionnaires concerning Restless Legs Syndrome(RLS)-symptoms and sleep quality will show the effect of iv-Iron supplementation on Restless Legs Syndrome(RLS)-symptoms during pregnancy.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

1. Pregnant women, singleton pregnancy, in the 3rd trimester
2. Iron Deficiency (Anaemia) defined as Serum Ferritin < 35ug/l with or without Hb < 11g/dl.
3. Fulfilling the 4 criteria of the International Restless Legs Study Group (IRLSS)

   * Uncomfortable and unpleasant sensations in the legs
   * An urge to move the legs due to this discomfort and worsening of the symptoms when resting
   * The unpleasant sensations are being relieved by movement such as walking or stretching
   * Worsening of the symptoms in the evening or night
4. RLS score > 20 (defined as modest to severe RLS symptoms) or RLS symptoms = 3 times per week
5. Patients = 18 years
6. Signed informed consent provided

Exclusion criteria: Criteria

1. Age < 18 years
2. Multiple pregnancy
3. Depression, psychiatric disease
4. Severe internal underlying disease, that causes fatigue and sleepiness and thus may confound the outcome measures
5. Abuse of alcohol, coffee or drugs
6. Medication (antipsychotics, antihistaminics, tricyclic or SSRI/SNRI antidepressants, L-Dopa, antidopaminergic medication, medium to strong opioids, antiepileptic medication).
7. RLS not due to iron deficiency: RLS secondary to other central nervous system disease or injury. Such disorders included peripheral neuropathy, neurodegenerative disorders and multiple sclerosis
8. RLS secondary to chronic kidney disease
9. Relevant chronic pain syndrome of the extremities other than RLS
10. Known proneness to allergic reactions
11. Known hypersensitivity to Ferric carboxymaltose
12. Relevant disorders of iron metabolism of other aetiology than iron deficiency (e.g. hemochromatosis, hemosiderosis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: = 50% reduction of RLS symptoms as measured by International Restless Legs Study Group (IRLSS) | 3 days, 7 days, 14 days, 28 days, and 60 days after iron infusion

SECONDARY OUTCOMES:
Reduction of Periodic Limb Movements in Sleep (PLMS) ≥50% as measured with actimetry | screening, 7 days, 14 days after iron infusion
Improvement of sleep according to the Pittsburgh Sleep Quality Questionnaire (PSQI) | screening, 7 days after iron infusion, 14 days post partum
Improvement of sleepiness using Epworth Sleepiness Scale (ESS) | screening, 7 days, 14 days, 28 days after iron infusion, 14 days post partum
Improvement of fatigue using Fatigue Severity Scale (FSS) | screening, 7 days, 14 days, 28 days after iron infusion, 14 days post partum
Safety of ferric carboxymaltose during pregnancy in the 3rd trimester | Day 1, Day 3, Day 7, Day 14, Day 28, 14 days pre partum, 14 days post partum
  Recording of adverse events
Parameters of the newborn baby (apgar, umbilical artery pH, weight, mode of delivery) | 8 weeeks

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Bassetti, Professor, Principal Investigator — University Hospital Zurich, Neurology; Claudio Bassetti, Professor, Principal Investigator — Neuroenter of Southern Switzerland, Ospedale Civico, Lugano
Locations (2):
- Switzerland (2):
  - University Hospital Zurich, Neurology, Zurich, Canton of Zurich
  - Neurocenter of Southern Switzerland, Ospedale Civico, Lugano, Canton Ticino